CLINICAL TRIAL: NCT05459415
Title: Reducing Excision Margins After Neoadjuvant Chemoimmunotherapy for HPV Negative Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma (REMATCH)
Brief Title: Reducing Excision Margins After Neoadjuvant Chemoimmunotherapy for HPV Negative Resectable Locally Advanced HNSCC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REMATCH2201
Record Dates: First submitted 2022-06-22; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-06

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Neoadjuvant Therapy; Resection Margin
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reducing Excision Margins (Experimental): In resectable HPV-negative locally advanced head and neck squamous cell carcinoma, 3 cycles of preoperative neoadjuvant chemotherapy combined with immunotherapy are proposed, in patients with significant tumor shrinkage (≥50%) as assessed by imaging, to conduct research on narrowing the scope of surgery, preserve the patient's organ function, improve or improve the quality of life, and achieve a curative effect that is not inferior to traditional radical surgery
  Interventions: Procedure: Reducing Excision Margins

INTERVENTIONS:
Procedure: Reducing Excision Margins — Reducing Excision Margins After Neoadjuvant Chemoimmunotherapy

SUMMARY:
This study aims to explore the 2-year DFS (disease-free survival) rate and organ retention rate and to explore the ORR, PCR rate, 2y-OS， and quality of life of patients.

DETAILED DESCRIPTION:
This study aims to explore the 2-year DFS (disease-free survival) rate and organ retention rate after AP chemotherapy combined with anti-PD-1 antibody neoadjuvant treatment for HPV negative operable locally advanced head and HNSCC, and to explore the ORR, PCR rate, 2y-OS, and quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18-70 years old, gender is unlimited;
2. Histological diagnosis of oral, oropharyngeal, hypopharyngeal, or laryngeal squamous cell carcinoma; preoperative evaluation can be surgical resection.
3. HPV negative evaluation criteria: P16 immunohistochemistry is negative, that is, p16 is less than 70% negative, and negative HPV FISH test shall prevail; locally advanced, defined as per the United States Joint Committee on Cancer [AJCC] guidelines: -HPV negative disease, III, IVa, IVb; no previous tumor treatment for head and neck squamous cell carcinoma;
4. According to the RECIST version 1.1 standard, With at least one evaluable target lesion;
5. the ECOG physical status is 0-1 points;
6. the main organ function is normal, That is, the following standards should meet: (1) routine blood inspection standards should meet: (no blood transfusion within 14 days) a. Hb 90g / L: b. ANC≥1.5x109/L; c. PLT 80x109 / L; (2) biochemical inspection should meet the following standards a.BIL <1.25 times the upper normal value limit (ULN); b.ALT and AST<2.5xULN; In case of liver metastases, Then, ALT and AST <5xULN: c. Serum Cr ULN, Endophytic creatinine clearance> 50ml / min (Cockcroft-Gaut formula);
7. Signed written informed consent prior to any test-related activity;
8. Investigators judged the ability to comply with the study protocol;
9. pregnancy test at screening (for fertile female patients) negative;
10. Fertility of male patients and female patients at risk of fertility and pregnancy must agree to the use of two contraceptive methods (at least one of which is considered efficient) throughout the study period. Unfertile women (i. e., meet one of at least the following criteria): -hysterectomy and/or bilateral oophorectomy with documented records; -medically confirmed ovarian function decline; -Postmenopausal status, defined as menopause for at least 12 consecutive months of menopause without other pathologic or physiologic reasons and confirmed by serum follicle-stimulating hormone (FSH) levels.
11. Patients who are willing and able to comply with visit schedules, treatment plans, laboratory tests, and other research procedures.12 A signed and dated informed consent indicates that the patient (or legal representative, if permitted by local guidelines/practice practices) has been informed of all relevant aspects of the study

Exclusion Criteria:

1. Previous immunotherapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibodies (including ipilimumab), or any other antibodies or drugs specifically targeted to the T cell co-stimulation or immune checkpoint pathway.
2. Major surgery for the first 4 weeks before enrollment;
3. People with a proven allergy to PD-1 antibody or its excipients;
4. Any active autoimmune disease or a history of autoimmune disease (e. g., Interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, reduced thyroid function (can be included after effective hormone replacement therapy): vitiligo or asthma in childhood, Asthmatic patients living in adults, either without any intervention and requiring medical intervention with bronchodilators, may be included);
5. Previous or concurrent cases of other malignancies (cured, Except for malignancies with cancer-free survival of more than 5 years, Such as skin basal cell carcinoma, cervical carcinoma in situ, and papillary thyroid carcinoma);
6. Heart clinical symptoms or diseases that cannot be controlled, For example: (1) heart failure of grade NYHAII or above (2) unstable heart pattern pain (3) myocardial infarction within 1 year (4) patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
7. Within 14 days before the administration of the study drug, Subjects who require systemic treatment with corticosteroids (> 10 mg/day, an efficacy dose of prednisone) or other immunosuppressants, In the absence of active autoimmune disease, Allow inhaled or topical use of steroids and adrenal hormone replacement with efficacy doses of prednisone> 10 mg/day；
8. Active infection requiring treatment;
9. Having an innate or acquired immune deficiency (e. g., an HIV-infected person), active hepatitis B (HBV-DNA 104 copy number/ml or 2000IU / ml), or hepatitis C (hepatitis C antibody positive, And HCV-RNA is above the lower limit of analysis);
10. Patients have received other oncology treatments before treatment;
11. Live vaccine within 4 weeks before the start of study treatment;
12. Known history of psychotropic substance abuse, alcohol or drug use;
13. Women during pregnancy or lactation;
14. Researchers judge, Subjects had other factors that could contribute to their forced termination of the study midway, If other serious diseases (including mental illness) require combined treatment, Laboratory examination values were seriously abnormal, Family or social factors, May affect the subject safety or trial data collection;
15. Patients considered not feasible for radical resection;
16. active tuberculosis;
17. Severe infections occurring within 4 weeks prior to initiation of study treatment (including but not limited to hospitalization, due to complications of infection, bacteremia or severe pneumonia);
18. Receiving systemic immune stimulation medication within 4 weeks before initiation of study treatment (including but not limited to interferon or interleukin-2 [IL-2]) or remaining in 5 drug half-lives (older of both).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-06-21 (Estimated); Study Completion 2027-06-21 (Estimated)

PRIMARY OUTCOMES:
DFS（disease-free survival） | 2 years
  2 years disease-free survival

SECONDARY OUTCOMES:
Organ retention rate | 2 years
  Organ retention rate

OTHER OUTCOMES:
ORR | 2 years
  tumor objective response rate
pCR | 2 years
  Pathologic Complete Response

CONTACTS AND LOCATIONS:
Overall Officials: kunyu Mr Yang, Doctor, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Zhanjie Zhang, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Winquist E, Agbassi C, Meyers BM, Yoo J, Chan KKW; Head and Neck Disease Site Group. Systemic therapy in the curative treatment of head-and-neck squamous cell cancer: Cancer Care Ontario clinical practice guideline. Curr Oncol. 2017 Apr;24(2):e157-e162. doi: 10.3747/co.24.3489. Epub 2017 Apr 27. PMID 28490940
- [Result] Szturz P, Wouters K, Kiyota N, Tahara M, Prabhash K, Noronha V, Castro A, Licitra L, Adelstein D, Vermorken JB. Weekly Low-Dose Versus Three-Weekly High-Dose Cisplatin for Concurrent Chemoradiation in Locoregionally Advanced Non-Nasopharyngeal Head and Neck Cancer: A Systematic Review and Meta-Analysis of Aggregate Data. Oncologist. 2017 Sep;22(9):1056-1066. doi: 10.1634/theoncologist.2017-0015. Epub 2017 May 22. PMID 28533474
- [Result] Lorch JH, Goloubeva O, Haddad RI, Cullen K, Sarlis N, Tishler R, Tan M, Fasciano J, Sammartino DE, Posner MR; TAX 324 Study Group. Induction chemotherapy with cisplatin and fluorouracil alone or in combination with docetaxel in locally advanced squamous-cell cancer of the head and neck: long-term results of the TAX 324 randomised phase 3 trial. Lancet Oncol. 2011 Feb;12(2):153-9. doi: 10.1016/S1470-2045(10)70279-5. Epub 2011 Jan 11. PMID 21233014
- [Result] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Result] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Result] Pasquali S, Chiarion-Sileni V, Rossi CR, Mocellin S. Immune checkpoint inhibitors and targeted therapies for metastatic melanoma: A network meta-analysis. Cancer Treat Rev. 2017 Mar;54:34-42. doi: 10.1016/j.ctrv.2017.01.006. Epub 2017 Feb 2. PMID 28189914
- [Result] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Result] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Result] Duray A, Demoulin S, Hubert P, Delvenne P, Saussez S. Immune suppression in head and neck cancers: a review. Clin Dev Immunol. 2010;2010:701657. doi: 10.1155/2010/701657. Epub 2011 Mar 10. PMID 21437225
- [Result] Ogino T, Shigyo H, Ishii H, Katayama A, Miyokawa N, Harabuchi Y, Ferrone S. HLA class I antigen down-regulation in primary laryngeal squamous cell carcinoma lesions as a poor prognostic marker. Cancer Res. 2006 Sep 15;66(18):9281-9. doi: 10.1158/0008-5472.CAN-06-0488. PMID 16982773
- [Result] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Result] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Result] Cloughesy TF, Mochizuki AY, Orpilla JR, Hugo W, Lee AH, Davidson TB, Wang AC, Ellingson BM, Rytlewski JA, Sanders CM, Kawaguchi ES, Du L, Li G, Yong WH, Gaffey SC, Cohen AL, Mellinghoff IK, Lee EQ, Reardon DA, O'Brien BJ, Butowski NA, Nghiemphu PL, Clarke JL, Arrillaga-Romany IC, Colman H, Kaley TJ, de Groot JF, Liau LM, Wen PY, Prins RM. Neoadjuvant anti-PD-1 immunotherapy promotes a survival benefit with intratumoral and systemic immune responses in recurrent glioblastoma. Nat Med. 2019 Mar;25(3):477-486. doi: 10.1038/s41591-018-0337-7. Epub 2019 Feb 11. PMID 30742122
- [Result] Pircher A, Gamerith G, Amann A, Reinold S, Popper H, Gachter A, Pall G, Woll E, Jamnig H, Gastl G, Wolf AM, Hilbe W, Wolf D. Neoadjuvant chemo-immunotherapy modifies CD4(+)CD25(+) regulatory T cells (Treg) in non-small cell lung cancer (NSCLC) patients. Lung Cancer. 2014 Jul;85(1):81-7. doi: 10.1016/j.lungcan.2014.04.001. Epub 2014 Apr 13. PMID 24780112
- [Result] Lacas B, Carmel A, Landais C, Wong SJ, Licitra L, Tobias JS, Burtness B, Ghi MG, Cohen EEW, Grau C, Wolf G, Hitt R, Corvo R, Budach V, Kumar S, Laskar SG, Mazeron JJ, Zhong LP, Dobrowsky W, Ghadjar P, Fallai C, Zakotnik B, Sharma A, Bensadoun RJ, Ruo Redda MG, Racadot S, Fountzilas G, Brizel D, Rovea P, Argiris A, Nagy ZT, Lee JW, Fortpied C, Harris J, Bourhis J, Auperin A, Blanchard P, Pignon JP; MACH-NC Collaborative Group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): An update on 107 randomized trials and 19,805 patients, on behalf of MACH-NC Group. Radiother Oncol. 2021 Mar;156:281-293. doi: 10.1016/j.radonc.2021.01.013. Epub 2021 Jan 27. PMID 33515668
- [Result] Cohen EE, Karrison TG, Kocherginsky M, Mueller J, Egan R, Huang CH, Brockstein BE, Agulnik MB, Mittal BB, Yunus F, Samant S, Raez LE, Mehra R, Kumar P, Ondrey F, Marchand P, Braegas B, Seiwert TY, Villaflor VM, Haraf DJ, Vokes EE. Phase III randomized trial of induction chemotherapy in patients with N2 or N3 locally advanced head and neck cancer. J Clin Oncol. 2014 Sep 1;32(25):2735-43. doi: 10.1200/JCO.2013.54.6309. Epub 2014 Jul 21. PMID 25049329

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT05459415/Prot_SAP_ICF_000.pdf